CLINICAL TRIAL: NCT02949063
Title: The Comfortable Cafeteria Program for Promoting Student Participation and Enjoyment: An Outcome Study
Brief Title: Creating a Comfortable Cafeteria: Staff and Student Feedback - Outcome Study (Cafeteria Prog)
Acronym: CCProgram
Status: Completed | Type: Observational
Sponsor: Mary Jane Karpinski (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Mary Jane Karpinski, Administrative Assistant, Office of Research Services, Cleveland State University
Organization: Cleveland State University (Other)
Other Study IDs: 29789-BAZ-HS; H027A130158-13A, CFDA 84.027A (Other Grant/Funding Number: Ohio Department of Education)
Record Dates: First submitted 2016-10-26; First posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: School Health Services
Keywords: school lunch; occupational therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Comfortable Cafeteria Program — 6-week program integrated into the cafeteria lunchtime to build capacity of supervisors and students to create a positive social and emotional atmosphere so that students can enjoy eating their lunch and socializing with peers.

SUMMARY:
A mixed methods design was used to explore the outcomes of a 6-week, occupational therapy-led Comfortable Cafeteria program designed to build capacity of cafeteria supervisors to create a positive mealtime environment so that all students can successfully participate in and enjoy their meal and socialization with peers.

DETAILED DESCRIPTION:
A mixed methods design was used to explore the outcomes of a 6-week, occupational therapy-led Comfortable Cafeteria program designed to build capacity of cafeteria supervisors to create a positive mealtime environment so that all students can successfully participate in and enjoy their meal and socialization with peers. Statistically significant improvements in pretest posttest visual analogue scale ratings of participation in and enjoyment for students with low and mid-range scores at the outset was found. Cafeteria supervisors demonstrated statistically significant improvements in perceptions of having the knowledge and skills to supervise and to encourage healthy eating based on pretest posttest ratings. Qualitative findings add further insight about the program suggesting that students learned prosocial values (e.g. being kind, helping others), supervisors actively encouraged positive social interaction, and occupational therapy practitioners enjoyed implementing the Comfortable Cafeteria program and recognized positive supervisor and student changes as a result of integrating services in the cafeteria.

ELIGIBILITY:
Inclusion Criteria:

* Students participating in lunch from a particular grade
* Cafeteria supervisors of those children
* Students with parental consent

Exclusion Criteria:

* Students who did not have parental consent

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 366 kindergarten through 4th grade students
  18 cafeteria supervisors
Sampling Method: Non-Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
students' participation during lunch | within 6 weeks
  Visual analogue scale

SECONDARY OUTCOMES:
survey of cafeteria supervisor's knowledge, beliefs and actions related to supervising students in the cafeteria | 6 weeks
  written pre and post-survey

CONTACTS AND LOCATIONS:
Overall Officials: Susan Bazyk, PhD, Principal Investigator — Cleveland State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bazyk S, Demirjian L, Horvath F, Doxsey L. The Comfortable Cafeteria Program for Promoting Student Participation and Enjoyment: An Outcome Study. Am J Occup Ther. 2018 May/Jun;72(3):7203205050p1-7203205050p9. doi: 10.5014/ajot.2018.025379. PMID 29689174
- See also: Comfortable Cafeteria program information is located on this website including instructions for implementation. — http://www.everymomentcounts.org